CLINICAL TRIAL: NCT03740217
Title: Comparison of the Relative Oral Bioavailability of GKT137831 Formulated in Capsules or in Tablets and Evaluation of the Potential Impact of Concomitant Food Intake on the Relative Bioavailability of GKT137831 in Healthy Male Subjects
Brief Title: Comparison of the Relative Oral Bioavailability of GKT137831 Formulated in Capsules or in Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calliditas Therapeutics AB (Industry)
Collaborators: Eurofins Optimed (Industry); York Bioanalytical Solution (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GSN000299
Record Dates: First submitted 2018-10-12; First posted 2018-11-14 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2019-01

CONDITIONS: Phase 1
MeSH Terms: interventions — setanaxib

STUDY DESIGN:
Intervention Model Description: Subject will be randomly allocated with different formulations of treatment or conditions (Fasting or Fed) during three periods (P1, P2 and P3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment A (Other): Single oral dose of 400 mg GKT137831 administered as 4 x 100 mg capsules in fasting conditions.
  Interventions: Drug: GKT137831
- Treatment B: (Other): Single oral dose of 400 mg GKT137831 administered as 1 x 400 mg tablets in fasting conditions.
  Interventions: Drug: GKT137831
- Treatment C (Other): Single oral dose of 400 mg GKT137831 administered as 1 x 400 mg tablets in fed conditions.
  Interventions: Drug: GKT137831

INTERVENTIONS:
Drug: GKT137831 — oral bioavailable small molecule that selectively inhibit NOX1 and NOX4
  Other Names: NOX1/4 inhibitor

SUMMARY:
The study will be a comparative oral bioavailability study between GKT137831 capsules and tablets, together with an assessment of the impact of concomitant food intake on the relative bioavailability of GKT137831 tablets.

This will be a randomized three-way open cross-over study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subject, aged 18 to 60 years inclusive;
2. Non-smoker subject or smoker of not more than 5 cigarettes a day ;
3. No history of alcohol or drug abuse
4. Body Mass Index (BMI) between 18 and 27 5 kg/m2 inclusive;
5. Considered as healthy after a comprehensive clinical assessment (detailed medical history and complete physical examination);
6. Signing a written informed consent prior to selection;

Exclusion Criteria:

1. Blood donation (including in the frame of a clinical study) within 2 months before administration;
2. General anaesthesia within 3 months before administration;
3. Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician;
4. Inability to abstain from intensive muscular effort;
5. No possibility of contact in case of emergency;
6. Any drug intake (except paracetamol) during the last month prior to the first administration;
7. History or presence of drug or alcohol abuse (alcohol consumption > 40 grams / day);
8. Excessive consumption of beverages with xanthine bases (> 4 cups or glasses / day);
9. Positive Hepatitis B surface (HBs) antigen or anti Hepatitis C Virus (HCV) antibody, or positive results for Human Immunodeficiency Virus (HIV) 1 or 2 tests;
10. Positive results of screening for drugs of abuse;
11. Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development;
12. Exclusion period of a previous study;
13. Administrative or legal supervision;

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Oral bioavailability (Fz) | 72 hours
  To compare the relative oral bioavailability GKT137831 formulated in capsules or in tablets in healthy male subjects.
Food effect on Oral bioavailability (Fz) | 72 hours
  To assess the impact of concomitant food intake on the relative bioavailability of GKT137831 after single oral dose administration of a 400 mg GKT137831 tablet in healthy male subjects.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 7 days
  To compare the safety and tolerability of single oral dose administration of 400 mg GKT137831 formulated in capsules or in tablets, and to evaluate the potential impact of concomitant food intake on the safety and tolerability of single oral dose administration of 400 mg GKT137831 tablet in healthy adult male subjects.
Oral bioavailability of GKT138184 | 72 hours
  To compare the relative oral bioavailability GKT138184 after oral administration of GKT137831 formulated in capsules or in tablets in healthy male subjects.
Food effect on oral bioavailability of GKT138184 | 72 hours
  To assess the impact of concomitant food intake on the relative bioavailability of GKT138184 after single oral dose administration of a 400 mg GKT137831 tablet in healthy male subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Yves DONAZZOLO, MD, Principal Investigator — Eurofins Optimed
Locations (1):
- Eurofins Optimed, Gières, France

IPD SHARING:
Plan to Share IPD: Undecided